CLINICAL TRIAL: NCT01850290
Title: Imaging Dopamine Function and Its Impact on Outcome After Traumatic Brain Injury (TBI)
Status: Completed | Type: Observational
Sponsor: Baylor Research Institute (Other)
Collaborators: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 012-277; H133A120098 (Other Grant/Funding Number: NIDRR)
Record Dates: First submitted 2013-05-07; First posted 2013-05-09 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Traumatic Brain Injury
Keywords: TBI
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dopamine Imaging

SUMMARY:
This study will examine resting dopamine function as well as dopamine response in the brain as it interacts with medicines normally prescribed to subacute Traumatic Brain Injury (TBI) patients.

ELIGIBILITY:
Inclusion Criteria:

* Non-penetrating TBI
* Age between 18-50 years old
* Admitted to a North Texas TBI Model Systems-affiliated rehabilitation facility within 16 weeks of injury
* Rated at Rancho VI Los Amigos Levels of Cognitive Functioning Scale of less than or equal to Stage V at the time of enrollment
* Disability Rating Scale total score >/= 7

Exclusion Criteria:

* Central Nervous System disorder resulting in functional disability predating TBI
* Documented diagnosis of disease processes impacted by the dopamine system (e.g., Parkinson's Disease, clinician diagnosed Attention Deficit Hyperactivity Disorder, substance abuse/dependence (excluding marijuana, alcohol, tobacco), or schizophrenia)
* Pre-injury use of dopaminergic pharmaceuticals (i.e., methylphenidate, amantadine, or dopamine receptor blockers such as olanzapine or quetiapine)
* Documented contraindication to use of methylphenidate including allergy
* Uncontrolled epilepsy
* Pregnant
* Medical condition not compatible with use of Methylphenidate
* Recent diagnosis or therapeutic study using radiopharmaceuticals
* Contraindications to the use of Ioflupane
* Allergic to Iodine

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Traumatic Brain Injury patients in Inpatient Rehabilitation
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in Disability Rating Scale | Baseline, 1 week, 2 weeks, 3 weeks, 4 weeks
  The primary outcome measure will be the change in Disability Rating Scale over 4 weeks. The Disability Rating Scale is a commonly used and reliable instrument for monitoring minor changes occurring throughout the course of a patient's recovery (Rappaport et al., 1982).

SECONDARY OUTCOMES:
John F Kennedy Coma Recovery Scale Revised | Baseline, 1 week, 2 weeks, 3 weeks, 4 weeks
Functional Independence Measure (FIM) | Baseline, 1 week, 2 weeks, 3 weeks, 4 weeks
Functional Assessment Measure (FAM) | Baseline, 1 week, 2 weeks, 3 weeks, 4 weeks
Orientation Log (O-Log) | Baseline, 1 week, 2 weeks, 3 weeks, 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shahid Shafi, MD, Principal Investigator — Baylor Research Institute; Devous Michael, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Baylor Research Institute, Dallas, Texas, United States